CLINICAL TRIAL: NCT06382038
Title: Smart Technology Facilitated Patient-centered Care for Patients With Pulmonary Thromboembolism：A Multicenter, Randomized Controlled Trial
Brief Title: Smart Technology Facilitated Patient-centered Care for Patients With Pulmonary Thromboembolism
Acronym: SmaPE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Navy General Hospital, Beijing (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: HZKY-PJ-2024-19
Record Dates: First submitted 2024-04-18; First posted 2024-04-24 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Venous Thromboembolism; Pulmonary Thromboembolisms; Digital Health
Keywords: Venous Thromboembolism; Pulmonary Thromboembolisms; Digital Health
MeSH Terms: conditions — Venous Thromboembolism; Pulmonary Embolism

STUDY DESIGN:
Intervention Model Description: This study is a multicenter, prospective, randomized controlled trial with a superiority design. Consecutively recruited patients with PTE will be randomly assigned in a 2:1 ratio to the interventive arm (mobile VTE application, mVTEA) and the usual care arm.
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- mVTEA Management Group (Experimental): Patients randomly assigned to the mVTEA management group will be discharged with mVTEA-assisted patient-centered PTE management.
  Interventions: Other: mobile venous thromboembolism application (mVTEA)
- Routine Management Group (No Intervention): Patients randomly assigned to the routine management group will be given routine post-discharge management in accordance with local clinical practice.

INTERVENTIONS:
Other: mobile venous thromboembolism application (mVTEA) — mVTEA will assist in the management of patients during the post-hospitalization follow-up phase. The mVTEA's doctor terminal automatically sends venous thromboembolism (VTE)-related health education materials in different frequencies and contents based on the patient's knowledge of VTE prevention and treatment, as well as their risk of thrombosis and bleeding during follow-up. In addition, thrombosis physicians on the mVTEA's doctor terminal can deliver health education to patients based on their condition. This can be done through the mVTEA doctor-patient communication module, which includes text, voice, and video communication.
  Arms: mVTEA Management Group

SUMMARY:
Smart technologies, such as wearable devices, mobile technologies, and artificial intelligence, are being investigated for use in health management. These technologies have the potential to be applied in disease pre-warning, decision-making support, health education, and healthcare maintenance. They are expected to address the challenges in managing thrombosis, improve access to high-quality medical resources in various regions, and enhance the development of a network for thrombosis rescue and treatment prevention.

The objective of this study is to evaluate the impact of mobile venous thromboembolism application (mVTEA) based patient-centered management of pulmonary thromboembolism (PTE) on the long-term outcome of PTE patients, in order to enhance clinical practice and establish a foundation of evidence for managing patients with PTE.

ELIGIBILITY:
Inclusion Criteria:

* Inpatients aged ≥18 years;
* （2）PTE confirmed through imaging examinations, meeting at least one of the following criteria: a.Newly diagnosed PTE during the current hospitalization; b. Prior PTE with imaging evidence of residual thrombus.
* Signed informed consent.

Exclusion Criteria:

* Previous PTE combined with CTEPH;
* Mental retardation or a combination of other serious illnesses that make them incapable of living on their own;
* Inability to use smartphones, computer tablets and other smart devices;
* Being pregnant or breastfeeding;
* Have participated in similar trials or are undergoing other clinical trials.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2972 (Estimated)
Dates: Start 2025-10-08 (Estimated); Primary Completion 2026-10-31 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
VTE-related composite event | At 1-year follow-up
  The primary outcome was the occurrence of VTE-related composite event at 1-year follow-up, which was defined as a composite of recurrent VTE, newly diagnosed deep vein thrombosis (DVT), chronic thromboembolic pulmonary hypertension (CTEPH), major bleeding, VTE-related rehospitalization, and all-cause death.

SECONDARY OUTCOMES:
VTE events | At 3, 6, 12, and 24-month follow-up
  VTE events will be documented at the 3, 6, 12, and 24-month follow-up after discharge. VTE events are categorized into two groups: recurrent VTE and newly diagnosed DVT.
  Recurrent VTE is defined as the appearance of new evidence of VTE after acute VTE has been treated in the acute phase (2 weeks) with significant clinical improvement in signs and symptoms. According to the time of VTE recurrence, it is further categorized into early VTE recurrence (within 3 months after the last VTE occurrence) and late VTE recurrence (more than 3 months after the last VTE occurrence).
  DVT that occurred for the first time after discharge during the study period is classified as newly diagnosed DVT.
Chronic thromboembolic pulmonary hypertension (CTEPH) | At 3, 6, 12, and 24-month follow-up
  The diagnosis of CTEPH will be documented at the 3, 6, 12, and 24-month follow-up.
Chronic thromboembolic pulmonary disease (CTEPD) | At 3, 6, 12, and 24-month follow-up
  The diagnosis of CTEPD will be documented at the 3, 6, 12, and 24-month follow-up after discharge.
Post-pulmonary embolism syndrome (PPES) | At 3, 6, 12, and 24-month follow-up
  The diagnosis of PPES will be documented at the 3, 6, 12, and 24-month follow-up after discharge
Major bleeding | At 3, 6, 12, and 24-month follow-up
  The major bleeding events as defined by the International Society on Thrombosis and Hemostasis (ISTH) will be documented at the 3, 6, 12, and 24-month follow-up after discharge.
VTE-related hospitalization | At 3, 6, 12, and 24-month follow-up
  Rehospitalization due to VTE recurrence, progression, or complications related to VTE treatment will be documented during the follow-up.
Death | At 3, 6, 12, and 24-month follow-up
  Death will be documented during the follow-up. It is categorized into all-cause death and PTE-related death. All-cause death is defined as death that occurs during the study period, regardless of cause. PTE-related death is defined as death that is unequivocally due to PTE.
Patient-Reported Outcome Events (PROs) | At 3, 6, 12, and 24-month follow-up
  PROs will be documented during the 3, 6, 12, and 24-month follow-up after discharge.
  PROs refer to information directly conveyed by patients themselves concerning their health status, symptoms, functional capacity, or adverse events related to treatment, without the need for interpretation or mediation by clinicians or other third parties.
Generic quality of life | At 6, 12, and 24-month follow-up
  Generic, non-disease-specific health-related quality of life (QoL) is assessed using the EuroQol 5-Dimension 5-Level (EQ-5D-5L) questionnaire and its corresponding visual analogue scale at 6, 12, and 24 months after discharge. Briefly, the EQ-5D-5L generates an overall index that ranges from 0 (lowest generic QoL) to 1 (highest generic QoL) and is calculated based on country-specific reference value sets. The EQ-5D-5L health index was calculated with the value set for China. The EuroQol visual analogue scale ranges from 0 to 100, with higher scores indicating better health.
Costs of management for healthcare staff | At 3, 6, and 12-month follow-up
  Costs of healthcare staff training (training duration × hourly wage), including training on standardized management of pulmonary embolism and the use of mVTEA; costs associated with post-discharge patient management by healthcare personnel (such as follow-up management, rehabilitation management, health counseling, and comorbidity management), calculated as (consultation time/re-hospitalization time × hourly wage); and development costs for mobile technology and intelligent algorithms.
Treatment costs for VTE-related patients | At 1-year follow-up
  Treatment costs for VTE-related patients within 12 months post-discharge: These include registration fees, diagnostic costs, and treatment expenses incurred during visits to community clinics, hospital emergency departments, or specialist outpatient clinics due to changes in PTE condition (such as VTE recurrence, newly diagnosed DVT, bleeding, CTEPH, CTEPD, or PPES). They also encompass diagnostic and treatment expenses during hospital admissions in community or specialist settings due to changes in PTE condition. Additionally, costs arising from routine VTE follow-ups (without any changes in VTE-related conditions) at community clinics, hospital emergency departments, or specialist outpatient clinics are included.
Treatment costs for non-VTE-related patients | At 3, 6, and 12-month follow-up
  Treatment costs for non-VTE-related patients within 12 months post-discharge: These comprise registration fees, diagnostic costs, and treatment expenses associated with visits to community clinics, hospital emergency departments, or specialist outpatient clinics for non-VTE-related conditions, as well as diagnostic and treatment expenses during hospital admissions in community or specialist settings for non-VTE-related diseases.
Anticoagulant adherence | At 3, 6, and 12-month follow-up
  Adherence would be assessed at months 3, 6, and 12 after discharge (defined as: the number of patients taking anticoagulants as prescribed/total number of patients at follow-up time point × 100%).
Probability of PTE progression | At 3, 6, and 12-month follow-up
  Clinical cure rate of PTE (defined as the numbers of patients without VTE recurrence, newly diagnosed DVT, bleeding, CTEPH, CTEPD, PPES, or all-cause mortality / total number of patients at the follow-up time point × 100% ); VTE (PTE/DVT) recurrence rate; incidence rate of newly diagnosed DVT; bleeding incidence rate; major bleeding incidence rate; non-major bleeding incidence rate; CTEPH incidence rate; CTEPD incidence rate; PPES incidence rate; all-cause mortality rate; PTE-related mortality rate would be collected.
Effectiveness evaluation | At 3, 6, and 12-month follow-up
  Quality-Adjusted Life Year(QALY) with EQ-5D-5L questionnaire would be investigated at 3, 6, and 12 months post-discharge and when the occurrence of VTE-related adverse events, including newly diagnosed DVT, bleeding, CTEPH, CTEPD, PPES, or all-cause mortality.

CONTACTS AND LOCATIONS:
Overall Officials: YU-TAO GUO, Doctor, Study Chair — Sixth Medical Center of Chinese PLA General Hospital
Locations (1):
- Sixth Medical Center of Chinese PLA General Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Valerio L, Mavromanoli AC, Barco S, Abele C, Becker D, Bruch L, Ewert R, Faehling M, Fistera D, Gerhardt F, Ghofrani HA, Grgic A, Grunig E, Halank M, Held M, Hobohm L, Hoeper MM, Klok FA, Lankeit M, Leuchte HH, Martin N, Mayer E, Meyer FJ, Neurohr C, Opitz C, Schmidt KH, Seyfarth HJ, Wachter R, Wilkens H, Wild PS, Konstantinides SV, Rosenkranz S; FOCUS Investigators. Chronic thromboembolic pulmonary hypertension and impairment after pulmonary embolism: the FOCUS study. Eur Heart J. 2022 Sep 21;43(36):3387-3398. doi: 10.1093/eurheartj/ehac206. PMID 35484821
- [Background] Schulman S, Angeras U, Bergqvist D, Eriksson B, Lassen MR, Fisher W; Subcommittee on Control of Anticoagulation of the Scientific and Standardization Committee of the International Society on Thrombosis and Haemostasis. Definition of major bleeding in clinical investigations of antihemostatic medicinal products in surgical patients. J Thromb Haemost. 2010 Jan;8(1):202-4. doi: 10.1111/j.1538-7836.2009.03678.x. Epub 2009 Oct 30. PMID 19878532